# Unstable Income, Rising Stress? The Effects of Income Instability on Psychological and Physiological Health

National Clinical Trial (NCT) Identified Number: Currently N/A

Principal Investigator: Heather Schofield

**Sponsor:** Cornell University

Grant Title: Unstable income, Rising Stress? The Effect of Income Instability on Psychological

and Physiological Health

**Grant Number\*:** Ro1AG076655

Funded by: National Institutes of Health (NIH) in the United States March 25, 2024

#### **INFORMED CONSENT - INFORMATION SHEET**

Title of Study: Economic uncertainty

#### Introduction

My name is Heather Schofield and I am the Principal Investigator for this study. I am working closely with Mr. Salifu Amadu and Mr. Abdul-Malik Abdul-Latif on this research.

Dr. Heather Schofield Assistant Professor, Cornell University 114 E Ave, Sage Hall 375; Ithaca NY 14853 +1 (617) 863-0726 hws44@cornell.edu

Mr.Salifu Amadu, Country Director. IPA Ghana. samadu@poverty-action.org

Mr. Abdul-Malik Abdul-Latif, Associate Research Manager. IPA Ghanaamlatif@poverty-action.org

# **Purpose and Nature of The Study**

To understand how employment and income might affect people's lives, this study will take place in this community and in other communities around this area. About 2,300 people will participate.

#### What Will We Ask You to Do if You Decide to Participate?

As part of the research study, you may be offered a job stitching bags. If you are offered the job, the amount of work may vary over time. Sometimes you may be offered more days of work; sometimes you may be offered fewer days. How much work is offered has nothing to do with you as a person. It is purely decided by a computer as we only have a certain number of days of work available.

You will be asked to work from home stitching bags and can choose your own hours.

Also, everyone will be asked to answer two different types of surveys. In one type of survey, someone will call you and ask you questions over the phone. There will be up to 6 calls. Each call will last about 20-30 minutes. In the other type of survey, someone will go to your home to interview you in person. There will be 2 of these interviews. Each interview will last no more than 3 hours. In these interviews, you will also be asked to provide a small sample of your hair which will allow us to measure a hormone which reflects stress. The hair will be discarded after it is tested.

#### **Risks & Benefits**

There are no serious anticipated risks associated with participation, just risks similar to those you face in your everyday life. There are also no benefits to you for participating.

#### **Duration**

Your participation in the study will last no more than 20 weeks. At most you will be offered work in 12 of these 20 weeks.

# Confidentiality

Your data will be kept confidential and stored at IPA Ghana. Your name and contact information will be stored separately from your survey answers and any other information about you, including a hair sample if you provide it.

# Outcome, Sharing of Anonymous Data, & Feedback

After the data is stripped of your personal information, it will be made publicly available for other researchers to study and for the funder of this study, the National Institutes of Health. Your personal information will be destroyed 3 years after the study ends. You will receive no feedback from the study.

## Compensation

You will be paid 12 GHS for each bag you sew. You will be paid 5GHS every time you complete a phone survey and 10 GHS for each in-person interview.

## **Costs**

None are anticipated.

#### **Participation & Withdrawal**

Your participation is completely voluntary. You may withdraw at any time without penalty. If you withdraw, you will keep the money you have earned until then. You may also choose to participate selectively. For example, you do not have to work all of the days that are offered. You can also choose to skip any survey questions you do not want to respond without penalty.

#### **Alternatives**

An alternative would be to not participate in this study.

#### **Funding**

This study is funded by the National Institutes of Health (NIH) in the United States.

# **Understanding**

Before you tell me if you want to participate, I'd like to ask you a few questions to make sure I explained you clearly and to give you a chance to ask any questions you may have.

- 1) If you decide you want to stop participating in the study, is this ok?
  - a) No, once you agree, you must continue
  - b) Yes, you can stop at any time without penalty
- 2) If you are offered a job, will you always work the same number of days?
  - a) No
  - b) Any other answer → reiterate that while many participants may receive work, not all will and the amount may vary over time.
- 3) How much are participants paid per bag sewn?
  - a) 12 GHS
  - b) Any other answer  $\rightarrow$  Participants are paid 12 GHS per bag produced.
- 4) How much do participants earn for each long survey they complete?
  - a) 10 GHS
  - b) Any other answer  $\rightarrow$  Participants are paid 10 GHS per long survey.

#### Provision of information and consent for participants

A copy of the Information Sheet and Consent Form will be given to you after it has been signed or thumb-printed for you to keep.

# Who to contact for further clarification/questions

Dr. Heather Schofield Assistant Professor, Cornell University +1 (617) 863-0726 hws44@cornell.edu

Ms. Sunny Liu Associate Research Manager-IPA Ghana sliu@poverty-action.org +233242343393

Ethics Review Committee (Note: The ERC Administrator should be contacted for ethical issues only)

Ghana Health Service

ethics.research@ghs.gov.gh

+233503539896

#### **Independent Contact**

Ethics Review Committee Ghana Health Service <a href="mailto:ethics.research@ghsmail.org">ethics.research@ghsmail.org</a>

+233503539896

#### **Informed Consent – Statement of Consent**

# PARTICIPANTS' STATEMENT

I voluntarily agree to be part of this research.

I acknowledge that I have read or have had the purpose and contents of the Participants' Information Sheet read and all questions satisfactorily explained to me in a language I understand (Dagbani). I fully understand the contents and any potential implications as well as my right to change my mind (i.e. withdraw from the research) even after I have signed this form.

| , - |
|---|
| Name of Participant |
| Participants' SignatureOR Thumb Print |
| Date: |
| SURVEYOR STATEMENT AND SIGNATURE |
| I was present when the purpose and contents of the Participant Information Sheet was read and explained satisfactorily to the participant in the language he/she understood (Dagbani). |
| I confirm that he/she was given the opportunity to ask questions/seek clarifications and same were duly answered to his/her satisfaction before voluntarily agreeing to be part of the research. |
| Name: |
| Signature Date: |